CLINICAL TRIAL: NCT03630484
Title: Comparison Between Ventilator Hyperinflation and Manual Rib Cage Compression: Randomized Crossover Trial
Brief Title: Ventilator Hyperinflation and Manual Rib Cage Compression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brazilian Institute of Higher Education of Censa (Other)
Responsible Party: Principal Investigator, Luciano Matos Chicayban, Principal Investigator, Brazilian Institute of Higher Education of Censa
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: VHI + Rib Cage Compression
Record Dates: First submitted 2018-08-06; First posted 2018-08-15 (Actual); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Pulmonary Atelectasis
Keywords: Ventilator Hyperinflation; Expiratory Rib Cage Compression; Physical Therapy; Mechanical Ventilation
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Expiratory Rib Cage Compression (Active Comparator): Expiratory rib cage compression was performed in 6 sets of 6 cycles, with 1 cycle interval. Ventilatory mode and parameters were maintained.
  Interventions: Other: Expiratory Rib Cage Compression
- Compression + Ventilator Hyperinflation (Active Comparator): Expiratory rib cage compression was performed in 6 sets of 6 cycles, with 1 cycle interval. Ventilator hyperinflation was performed by increasing the inspiratory pressure to every 5 cmH2O until the total pressure reached 40 cmH2O, remaining the same.
  Interventions: Other: Compression + Ventilator Hyperinflation

INTERVENTIONS:
Other: Expiratory Rib Cage Compression — Compression was performed in 6 sets of 6 cycles, with 1 cycle interval. Ventilatory mode and parameters were maintained.
  Arms: Expiratory Rib Cage Compression
Other: Compression + Ventilator Hyperinflation — Mechanical ventilator hyperinflation was performed by increasing the inspiratory pressure to every 5 cmH2O until the total pressure reached 40 cmH2O, remaining the same. In Expiratory Rib Cage Compression associated with ventilator hyperinflation, thoracic compression maneuver was performed at the end of inspiration, at the exact moment of cycling.
  Arms: Compression + Ventilator Hyperinflation

SUMMARY:
This is a randomized crossover trial to evaluate the effects of thoracic compression applied alone or in association with hyperinflation maneuver with the ventilator. In addition, the mobilized volume and peak expiratory flow resulting from both maneuvers will be evaluated.

DETAILED DESCRIPTION:
Ventilator hyperinflation is widely used in hypersecretive patients. It consists of increasing alveolar ventilation by facilitating the coughing mechanism so that the secretions of the peripheral airways are mobilized into the central airways so that they can be removed by tracheal aspiration or cough. Thoracic compression consists of manually compressing the rib cage during expiration, in order to increase expiratory flow, mobilize and remove pulmonary secretions. A randomized crossover clinical trial was performed with 30 patients submitted to isolated compression or associated with ventilator hyperinflation, with a 6 hour interval. Patients were evaluated through compliance and resistance of the respiratory system.

ELIGIBILITY:
Inclusion Criteria:

* patients under mechanical ventilation
* diagnosis of pulmonary infection
* hypersecretive

Exclusion Criteria:

* haemodynamic instability (heart rate > 130 bpm and mean arterial pressure < 60 mmHg)
* acute bronchospasm
* acute respiratory distress syndrome
* untreated pneumothorax

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-11-28 (Actual); Primary Completion 2014-12-05 (Actual); Study Completion 2017-07-11 (Actual)

PRIMARY OUTCOMES:
Static compliance of respiratory system | Baseline (before), immediately after ventilator hyperinflation or rib cage compression and five minutes after aspiration
  Compliance was assessed through the occlusion maneuver at the end of inspiration, considering tidal volume, plateau pressure and PEEP. Three measurements were taken at each moment, the mean being used.
Total Resistance of respiratory system | Baseline (before), immediately after ventilator hyperinflation or rib cage compression and five minutes after aspiration
  The total resistance of the respiratory system was evaluated through the occlusion maneuver at the end of the inspiration, considering the resistive pressure, measured by the difference between the maximum plateau pressure. Three measurements were taken at each moment, the mean being used.
Airway Resistance | Baseline (before), immediately after ventilator hyperinflation or rib cage compression and five minutes after aspiration
  The airway resistance was assessed by means of the occlusion maneuver at the end of the inspiration, considering the rapid fall of the pressure immediately after the occlusion, measured by the difference between the maximum pressure and P1. Three measurements were taken at each moment, the mean being used.
Peak expiratory flow | Baseline (before), immediately after ventilator hyperinflation or rib cage compression and five minutes after aspiration
  The peak expiratory flow was evaluated through passive expiration, being considered the greatest value of the flow in the expiratory phase.

CONTACTS AND LOCATIONS:
Overall Officials: LUCIANO M CHICAYBAN, MSc, Principal Investigator — Brazilian Institute of Higher Education of Censa

IPD SHARING:
Plan to Share IPD: No